CLINICAL TRIAL: NCT07131254
Title: A Clinical Study Evaluating the Safety and Efficacy of GT719 Universal Cell Injection in Adult Participants With Relapsed/Refractory CD19-positive B-cell Malignant Hematological Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Ganzhou City People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-001
Record Dates: First submitted 2025-06-26; First posted 2025-08-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hematological Malignancy (Leukemia- Lymphoma)
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: GT719 Injection

INTERVENTIONS:
Biological: GT719 Injection — GT719 Injection

SUMMARY:
This study is a prospective single-arm open-label clinical trial, including dose escalation and expansion phase, aims to evaluate the safety, efficacy, and cellular pharmacokinetics of GT719 Injection in relapsed/refractory CD19 positive adult B-cell non Hodgkin lymphoma (B-NHL) and B-acute lymphoblastic leukemia (B-ALL) patients. A total of 34 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily enrolled in the study, signed an informed consent form, willing and able to comply with the study protocol.
* 2. Aged 18 to 75 years (inclusive), regardless of gender.
* 3. Participants with refractory or relapsed acute B-cell lymphoblastic leukemia or B-cell lymphoma diagnosed according to the WHO 2016 classification.
* 4. CD19 positivity confirmed by flow cytometry and/or histopathology.
* 5. Eastern Collaborative Oncology Group (ECOG) physical fitness status score of 0 or 1.
* 6. Expected survival period > 12 weeks;
* 7. For any prior systemic therapy (excluding immune checkpoint inhibitors), at least 2 weeks or 5 half-lives (whichever is shorter) must have elapsed before the participant is scheduled to receive the study treatment. For any prior treatment with immune checkpoint inhibitors (such as anti-PD-1 or anti-PD-L1 monoclonal antibodies like Pembrolizumab, OX40 agonists, 4-1BB agonists, etc.), at least 3 half-lives or 28 days (whichever is shorter) must have passed before the participant is scheduled to receive the study treatment.
* 8. Toxicities caused by prior treatments must be stable and resolved to grade ≤ 1, excluding clinically insignificant toxicities such as alopecia.
* 9. Have adequate renal, hepatic, pulmonary, and cardiac functions, defined as follows:

  1. . Creatinine Clearance (estimated by the Cockcroft-Gault formula) ≥ 60 mL/min;
  2. . Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 times the Upper Limit of Normal (ULN);
  3. . Total bilirubin ≤ 1.5 mg/dl, excluding participants with Gilbert syndrome;
  4. . Cardiac ejection fraction ≥ 50%, no signs of pericardial effusion detected by Echocardiography (ECHO), and no clinically significant abnormalities found on Electrocardiogram (ECG);
  5. . No clinically significant pleural effusion;
  6. . Baseline oxygen saturation > 92% when measured under room air conditions.
* 10. Female participants of childbearing potential must have a negative result from a serum or urine pregnancy test. Females who have undergone surgical sterilization or been postmenopausal for at least 2 years are not considered to be of childbearing potential. They must agree to use highly effective and reliable contraceptive methods for 1 year after receiving the study treatment, and are strictly prohibited from donating oocytes within 1 year after the infusion of the study treatment during the study period.
* 11. Male participants who have active sexual life with females of childbearing potential must agree to use highly effective and reliable contraceptive methods for 1 year after receiving the study treatment. All male participants are strictly prohibited from donating sperm within 1 year after the infusion of the study treatment during the study period.

Exclusion Criteria:

* 1. Participants with a history of central nervous system (CNS) leukemia/lymphoma, or those with CNS leukemia/lymphoma shown by magnetic resonance imaging (MRI) or positron emission tomography-computed tomography (PET-CT) intracranial imaging during the screening period, or those with detected malignant cells in cerebrospinal fluid or brain metastases.
* 2. History of testicular leukemia/lymphoma, and imaging examinations during the screening period suggest active testicular leukemia/lymphoma.
* 3. History of other untreated malignant tumors within the past 5 years or concurrent with the current disease, excluding adequately treated carcinoma in situ of the cervix, localized cutaneous squamous cell carcinoma, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or ≤T1 urothelial carcinoma. Participants with prostate cancer undergoing active surveillance are eligible for this study;
* 4. Hematopoietic stem cell transplantation with curative intent performed within 6 weeks prior to the planned infusion of GT719 cells;
* 5. For participants with a history of hematopoietic stem cell transplantation, ≤6 months have elapsed since they received allogeneic hematopoietic stem cell transplantation;
* 6. History of CD19 CAR-T/NK therapy (except for participants who have received GT719 and are eligible for retreatment);
* 7. Received systemic glucocorticoid drugs within 7 days before cell infusion, except inhaled glucocorticoids.
* 8. History of allergic reactions to any components of the drugs intended for use in the study (including but not limited to the study drug GT719 cell infusion preparation, cyclophosphamide, and fludarabine).
* 9. Presence or suspicion of uncontrolled fungal, bacterial, viral, or other infections, or infections requiring management with intravenous (IV) antimicrobial agents;
* 10. Positive results for any of the following tests: Human Immunodeficiency Virus (HIV) antibody, Treponema pallidum antibody, Cytomegalovirus (CMV) IgM, Epstein-Barr Virus (EBV) IgM;
* 11. Active hepatitis B and/or active hepatitis C (HCV RNA positive); participants who are positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (anti-HBc) but with HBV-DNA levels within the normal range may be included;
* 12. Presence of any indwelling lines or drainage catheters (e.g., percutaneous nephrostomy tubes, indwelling Foley catheters, biliary drainage tubes, or pleural/peritoneal/pericardial catheters). Dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are permitted;
* 13. Presence or history of central nervous system (CNS) disorders, such as seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the CNS;
* 14. Participants with lymphoma involvement of the cardiac atria or ventricles.
* 15. Presence of any of the following within 6 months prior to signing the informed consent form: uncontrolled congestive heart failure (New York Heart Association Class III-IV, see Appendix III), angina pectoris, myocardial infarction, cardiomyopathy, stroke (excluding lacunar infarction), coronary/peripheral artery bypass surgery, clinically significant arrhythmias (as judged by the investigator) including but not limited to ventricular arrhythmias, significantly prolonged QT interval (QTc ≥500 ms corrected by the Bazett's method, as specifically judged by the investigator), poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg), poorly controlled diabetes mellitus, pulmonary embolism, diffuse pulmonary lesions, impaired pulmonary function, or any medical condition deemed by the investigator to be unsuitable for participation in this clinical study;
* 16. Participants for whom urgent treatment is expected or likely to be required within 6 weeks due to ongoing or impending tumor emergencies (e.g., tumor mass effect, tumor lysis syndrome);
* 17. Primary immunodeficiency.
* 18. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to enrollment, requiring systemic anticoagulant therapy;
* 19. Any medical condition that may interfere with the assessment of the safety or efficacy of the study treatment;
* 20. Vaccination with live attenuated vaccines or mRNA vaccines within 8 weeks prior to lymphodepleting conditioning, or inactivated vaccines within 4 weeks prior;
* 21. Females of childbearing potential who are pregnant or breastfeeding. Females who have undergone sterilization surgery or been postmenopausal for at least 2 years are not considered to be of childbearing potential;
* 22. Male and female participants who are unwilling to use contraception from the time of informed consent until 6 months after the completion of treatment.
* 23. Participants who, in the judgment of the investigator, are unlikely to complete all protocol-required study visits or procedures, including follow-up, or to comply with the requirements of study participation;
* 24. History of autoimmune diseases within the past 2 years that have caused end-organ damage or required systemic immunosuppressive agents/systemic disease-modifying agents (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 28 days
  Incidence and severity of Adverse events (AEs) occurring after infusion and their proportion
Proportion of participants experiencing dose limiting toxicity | 28 days
  Proportion of participants experiencing dose limiting toxicity (DLT) within 28 days after cell infusion

SECONDARY OUTCOMES:
overall response rate (ORR) | 3 months
  3 months overall response rate (ORR)
Best Overall Response（BOR） | 3 months
  3 months Best Overall Response（BOR）
Duration of Response（DOR） | 3 months
  3 months Duration of Response（DOR）
Progression-Free Survival（PFS） | 3 months
  3 months Progression-Free Survival（PFS）
Overall Survival（OS） | 3 months
  3 months Overall Survival（OS）
Time to Maximum Expansion of Infused Cells (Tmax) | From the time of infusion up to Month 3
  The time point at which the concentration of infused cells in peripheral blood reaches the peak level following product infusion, measured by flow cytometry
Peak Expansion Level of Infused Cells (Cmax) | From the time of infusion up to Month 3
  The maximum copy number or cell count of infused cells in peripheral blood after infusion, measured by flow cytometry
Area Under the Curve of Infused Cells (AUC) | From the time of infusion up to Month 3
  The area under the concentration-time curve of infused cells in peripheral blood from the time of infusion to the evaluation endpoint, reflecting the total exposure of cells in vivo
In Vivo Survival Time of Infused Cells | From the time of infusion up to Month 12
  The duration during which infused cells remain detectable in peripheral blood, defined as the time point when the cell concentration drops to the lower limit of detection

OTHER OUTCOMES:
Peripheral white blood cell count | From the time of infusion up to Month 3
  The measured total count of white blood cells in peripheral blood
Changes in peripheral white blood cell differential | From the time of infusion up to Month 3
  The dynamic changes in the quantity and proportion of various types of white blood cells in peripheral blood over time
Phenotypic changes of GT719 cells and other NKT cells | From the time of infusion up to Month 3
  Detect the dynamic changes in cell surface marker expression, morphological characteristics and function-related phenotypic features of GT719 cells and other natural killer T (NKT) cells
Changes in inflammatory factors in peripheral blood over different treatment time periods | From the time of infusion up to Month 3
  Dynamically monitor the concentration fluctuations of various inflammatory factors in peripheral blood during different treatment time periods
Anti-Drug Antibody (ADA) Testing | From the time of infusion up to Month 3
  Positive rate of detectable anti-CAR antibodies in serum at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- Ganzhou City People's Hospital, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No